CLINICAL TRIAL: NCT00999336
Title: Pharmacokinetics, Pharmacodynamics, and Tolerability of Betrixaban Administered Orally in Subjects With Normal and Reduced Renal Function.
Brief Title: A Study to Determine the Pharmacokinetics, Pharmacodynamics, and Tolerabiltiy of Betrixaban in Patients With Mild, Moderate, and Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-016
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2022-10

CONDITIONS: Renal Impairment
Keywords: Betrixaban; Renal impairment; Healthy; Kidney dysfunction
MeSH Terms: conditions — Renal Insufficiency | interventions — betrixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group H (Active Comparator): Healthy subjects matched to the renal impairment groups
  Interventions: Drug: Betrixaban
- Group A (Experimental): Patients with mild renal impairment
  Interventions: Drug: Betrixaban
- Group B (Experimental): Patients with moderate renal impairment
  Interventions: Drug: Betrixaban
- Group C (Experimental): Patients with severe renal impairment
  Interventions: Drug: Betrixaban

INTERVENTIONS:
Drug: Betrixaban — 80 mg betrixaban qd for 8 days

SUMMARY:
The purpose of the study is to compare the pharmacokinetics, pharmacodynamics, and tolerability of betrixaban in patients with mild, moderate, and severe renal impairment to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign the written informed consent.
* Subjects should have either normal renal function or have stable renal disease

Exclusion Criteria:

* Subjects require dialysis
* Evidence of active bleeding or bleeding disorder
* Unstable or clinically significant other disorders such as respiratory, hepatic, metabolic, psychiatric or gastrointestinal disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-07-31 (Actual); Primary Completion 2010-02-28 (Actual); Study Completion 2010-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- APEX GmbH, Munich, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 32 eligible participants were enrolled into 1 of 4 groups (8 participants per group) at screening according to the estimated glomerular filtration rate (eGFR).
Pre-assignment Details: Criteria based on age, gender, and weight were planned in order to match participants in the renal function groups and to ensure that renal function groups were comparable to each other.
Groups:
- Normal Renal Function: Participants with normal renal function according to the eGFR.
- Mild Renal Impairment: Participants with mild renal impairment according to the eGFR.
- Moderate Renal Impairment: Participants with moderate renal impairment according to the eGFR.
- Severe Renal Impairment: Participants with severe renal impairment according to the eGFR.
Period: Overall Study
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11.1) | 66 (6.2) | 69 (9.3) | 61 (12.1) | 64 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 1 | 11
  Male | 5 | 4 | 5 | 7 | 21
Race/Ethnicity, Customized [Number; unit: participants] — Population of participants based on their race.
  participants
    White | 8 | 8 | 8 | 8 | 32
Race/Ethnicity, Customized [Number; unit: participants] — Population of participants based on their ethnicity.
  participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 8 | 8 | 8 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Area Under The Plasma Concentration-Time Curve From Time Zero To 24 Hours (AUC0-24) Postdose Of Oral Doses Of Betrixaban On Day 8
Description: Blood and urine samples for pharmacokinetic analysis were collected and determined from the plasma and urine concentrations of betrixaban using non-compartmental procedures in WinNonlin Enterprise Version 5.2.
  Results were reported in nanogram multiplied by hour per milliliter (ng*h/mL).
Time Frame: Predose up to 168 hours postdose
Population: All participants with varying degrees of renal function who received the study intervention.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*h/mL | 437 (237) | 807 (254) | 1033 (549) | 995 (445)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; Test type: Other — Geometric least squares means, ratios, and confidence intervals (CIs) were estimated from an analysis of covariance (ANCOVA) of natural log transformed values; Ratio = 1.89, 90% CI 2-sided [1.18 to 3.03] — Statistical comparison of AUC0-24 on Day 8 for participants grouped using 186 as a multiplier in the Modified Diet in Renal Disease Study Group (MDRD) equation
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 2.27, 90% CI 2-sided [1.43 to 3.59] — Statistical comparison of AUC0-24 on Day 8 for participants grouped using 186 as multiplier in the MDRD equation
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 2.63, 90% CI 2-sided [1.71 to 4.06] — Statistical comparison of AUC0-24 on Day 8 for participants grouped using 186 as multiplier in the MDRD equation
Statistical Analysis 4: Comparison: Mild Renal Impairment vs Severe Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 1.39, 90% CI 2-sided [0.888 to 2.18] — Statistical comparison of AUC0-24 on Day 8 for participants grouped using 186 as multiplier in the MDRD equation
Statistical Analysis 5: Comparison: Normal Renal Function vs Mild Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 1.94, 90% CI 2-sided [1.14 to 3.31] — Statistical comparison of AUC0-24 on Day 8 for participants grouped using 175 as multiplier in the MDRD equation
Statistical Analysis 6: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 2.44, 90% CI 2-sided [1.41 to 4.22] — Statistical comparison of AUC0-24 on Day 8 for participants grouped using 175 as multiplier in the MDRD equation
Statistical Analysis 7: Comparison: Normal Renal Function vs Severe Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 2.86, 90% CI 2-sided [1.74 to 4.7] — Statistical comparison of AUC0-24 on Day 8 for participants grouped using 175 as multiplier in the MDRD equation
Statistical Analysis 8: Comparison: Mild Renal Impairment vs Severe Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 1.47, 90% CI 2-sided [0.944 to 2.3] — Statistical comparison of AUC0-24 on Day 8 for participants grouped using 175 as multiplier in the MDRD equation

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) Following Administration Of Oral Doses Of Betrixaban On Day 8
Description: Blood and urine samples for pharmacokinetic analysis were collected and determined from the plasma and urine concentrations of betrixaban using non-compartmental procedures in WinNonlin Enterprise Version 5.2.
  Results were reported in nanogram per milliliter (ng/mL).
Time Frame: Predose, up to 168 hours postdose
Population: All participants with varying degrees of renal function who received the study intervention.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL | 44.0 (24.4) | 84.3 (37.0) | 108 (59.1) | 104 (58.0)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 1.88, 90% CI 2-sided [1.05 to 3.35] — Statistical comparison of Cmax on Day 8 for participants grouped using 186 as multiplier in the MDRD equation
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 2.32, 90% CI 2-sided [1.32 to 4.07] — Statistical comparison of Cmax on Day 8 for participants grouped using 186 as multiplier in the MDRD equation
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 2.52, 90% CI 2-sided [1.48 to 4.29] — Statistical comparison of Cmax on Day 8 for participants grouped using 186 as multiplier in the MDRD equation
Statistical Analysis 4: Comparison: Mild Renal Impairment vs Severe Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 1.34, 90% CI 2-sided [0.772 to 2.32] — Statistical comparison of Cmax on Day 8 for participants grouped using 186 as multiplier in the MDRD equation
Statistical Analysis 5: Comparison: Normal Renal Function vs Mild Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 1.96, 90% CI 2-sided [1.01 to 3.78] — Statistical comparison of Cmax on Day 8 for participants grouped using 175 as multiplier in the MDRD equation
Statistical Analysis 6: Comparison: Normal Renal Function vs Moderate Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 2.38, 90% CI 2-sided [1.21 to 4.67] — Statistical comparison of Cmax on Day 8 for participants grouped using 175 as multiplier in the MDRD equation
Statistical Analysis 7: Comparison: Normal Renal Function vs Severe Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 2.69, 90% CI 2-sided [1.46 to 4.96] — Statistical comparison of Cmax on Day 8 for participants grouped using 175 as multiplier in the MDRD equation
Statistical Analysis 8: Comparison: Mild Renal Impairment vs Severe Renal Impairment; Test type: Other — Geometric least squares means, ratios, and CIs were estimated from an ANCOVA of natural log transformed values; Ratio = 1.37, 90% CI 2-sided [0.793 to 2.38] — Statistical comparison of Cmax on Day 8 for participants grouped using 175 as multiplier in the MDRD equation

3. Primary Outcome: Plasma Terminal Elimination Half-Life (T½) Following Administration Of Oral Doses Of Betrixaban On Day 8
Description: Blood and urine samples for pharmacokinetic analysis were collected and determined from the plasma and urine concentrations of betrixaban using non-compartmental procedures in WinNonlin Enterprise Version 5.2.
  Harmonic mean and Jackknife standard deviation was used to report this outcome and results were reported in hour.
Time Frame: Predose, up to 168 hours postdose
Population: All participants with varying degrees of renal function who received the study intervention.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour | 54.4 (9.20) | 56.0 (5.09) | 60.7 (8.17) | 55.6 (5.19)

4. Primary Outcome: Total Plasma Clearance (CL/F) Following Administration Of Oral Doses Of Betrixaban On Day 8
Description: Blood and urine samples for pharmacokinetic analysis were collected and determined from the plasma and urine concentrations of betrixaban using non-compartmental procedures in WinNonlin Enterprise Version 5.2.
  Results were reported in milliliter per minute (mL/min).
Time Frame: Predose, up to 168 hours postdose
Population: All participants with varying degrees of renal function who received the study intervention.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
mL/min | 4042 (2376) | 1815 (623) | 1887 (1468) | 1715 (1052)

5. Primary Outcome: Volume Of Distribution During The Terminal Phase (Vz/F) Following Administration Of Oral Doses Of Betrixaban On Day 8
Description: Blood and urine samples for pharmacokinetic analysis were collected and determined from the plasma and urine concentrations of betrixaban using non-compartmental procedures in WinNonlin Enterprise Version 5.2.
  Results were reported in liter.
Time Frame: Predose, up to 168 hours postdose
Population: All participants with varying degrees of renal function who received the study intervention.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
liter | 20128 (13391) | 8795 (2780) | 9518 (6183) | 9562 (6132)

6. Primary Outcome: Percentage Of Dose Excreted In Urine From 0-24 (fe0-24) Postdose Of Oral Doses Of Betrixaban On Day 8
Description: Blood and urine samples for pharmacokinetic analysis were collected and determined from the plasma and urine concentrations of betrixaban using non-compartmental procedures in WinNonlin Enterprise Version 5.2.
  Results were reported in percentage.
Time Frame: Predose, up to 24 hours postdose
Population: All participants with varying degrees of renal function who received the study intervention.
Measure: Mean (Standard Deviation); unit: percentage of excreted dose
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
percentage of excreted dose | 5.07 (2.32) | 5.40 (2.24) | 5.04 (2.38) | 2.72 (1.02)

7. Primary Outcome: Percentage Of Betrixaban Bound To Plasma Proteins On Day 8
Description: Blood samples were collected for measurement of plasma protein binding for betrixaban for all participants. Results of protein binding assays were summarized by sample time and eGFR group. Results were reported in percent (%).
Time Frame: 4 hours Postdose at Day 8
Population: All participants with varying degrees of renal function who received the study intervention.
Measure: Mean (Standard Deviation); unit: percentage of bound betrixaban
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
percentage of bound betrixaban | 58.6 (2.76) | 61.3 (1.86) | 59.4 (3.05) | 59.9 (3.62)

8. Primary Outcome: Thrombin Generation Following Administration Of Oral Doses Of Betrixaban On Day 8
Description: Blood samples were collected at the protocol-specified time points. Plasma samples were assayed for measurement of thrombin generation for all participants.
Time Frame: Day 1: predose; Day 8: 2, 3, 4, 8, 24, and 48 hours postdose
Population: All participants with varying degrees of renal function who received the study intervention.
Measure: Mean (Standard Error); unit: relative fluorescence units (RFU)
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
relative fluorescence units (RFU)
  Day 1 Predose | 12494 (2256.4) | 14168 (3387.2) | 11833 (3283.1) | 10021 (6034.7)
  Day 8 2 h | 6359 (2819.6) | 4484 (1411.4) | 4873 (1466.4) | 4773 (2059.1)
  Day 8 3 h | 6611 (1544.6) | 5356 (1632.2) | 5098 (1850.4) | 5547 (2994.4)
  Day 8 4 h | 6899 (1528.6) | 5103 (1406.7) | 6216 (3092.5) | 6154 (2818.6)
  Day 8 8 h | 9716 (1386.6) | 8789 (2923.8) | 7907 (2851.0) | 7482 (1959.3)
  Day 8 24 h: number analyzed (Participants) | 8 | 8 | 7 | 8
  Day 8 24 h | 8616 (2336.2) | 5870 (2205.7) | 7386 (1275.8) | 8013 (2710.4)
  Day 8 48 h | 12233 (3872.4) | 8350 (2863.9) | 8119 (1742.7) | 8485 (2858.0)

9. Primary Outcome: Anti-Factor Xa (fXa) Activity Following Administration Of Oral Doses Of Betrixaban On Day 8
Description: Blood samples were collected at the protocol-specified time points. Plasma samples were assayed for measurement of anti-fXa activity at baseline and steady state for all participants.
  Results were reported in international units per milliliter (IU/mL).
Time Frame: Day 8: 2, 3, 4, 8, 24, and 48 hours postdose
Population: All participants with varying degrees of renal function who received the study intervention.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
IU/mL
  Day 8 2 h: number analyzed (Participants) | 8 | 8 | 7 | 7
  Day 8 2 h | 0.18 (0.113) | 0.36 (0.293) | 0.48 (0.352) | 0.44 (0.237)
  Day 8 3 h: number analyzed (Participants) | 7 | 8 | 8 | 8
  Day 8 3 h | 0.27 (0.302) | 0.40 (0.163) | 0.60 (0.393) | 0.77 (0.453)
  Day 8 4 h: number analyzed (Participants) | 7 | 7 | 8 | 8
  Day 8 4 h | 0.22 (0.302) | 0.33 (0.116) | 0.58 (0.381) | 0.58 (0.310)
  Day 8 8 h | 0.10 (0.066) | 0.18 (0.070) | 0.32 (0.245) | 0.30 (0.276)
  Day 8 24 h: number analyzed (Participants) | 7 | 7 | 7 | 8
  Day 8 24 h | 0.06 (0.054) | 0.13 (0.056) | 0.18 (0.138) | 0.18 (0.123)
  Day 8 48 h: number analyzed (Participants) | 8 | 7 | 8 | 8
  Day 8 48 h | NA (NA) — Here, 'NA' signifies that the data was below the limit of quantification (BLQ) (0.1 IU/mL). | 0.08 (0.032) | 0.13 (0.082) | 0.12 (0.092)

ADVERSE EVENTS:
Time Frame: Day 1 through up to Day 12
Groups:
- Normal Renal Function: Participants with normal renal function according to the estimated eGFR.
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 1/8
Other Adverse Events (participants affected / at risk) | 5/8 | 3/8 | 5/8 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Renal Function (N=8) | Mild Renal Impairment (N=8) | Moderate Renal Impairment (N=8) | Severe Renal Impairment (N=8)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Renal Function (N=8) | Mild Renal Impairment (N=8) | Moderate Renal Impairment (N=8) | Severe Renal Impairment (N=8)
Gingival Bleeding (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes